CLINICAL TRIAL: NCT01365676
Title: Phase 3 Study Efficacy and Tolerance: The Use of 2 Phytomedicines in Association GAMALINE® 900mg + HIPERICIN® 300mg for the Treatment of Pre-Menstrual Syndrome (PMS) and Vasomotor Symptoms
Brief Title: GAMALINE®+HIPERICIN® for PMS Treatment and Vasomotor Symptoms
Acronym: 657/10UFCSPA
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Phytopharm Consulting Brazil (Network)
Collaborators: Herbarium Laboratorio Botanico Ltda (Industry); Federal University of Health Science of Porto Alegre (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: GAM+HIP
Record Dates: First submitted 2011-05-26; First posted 2011-06-03 (Estimated); Last update posted 2011-12-06 (Estimated); Status verified 2011-12

CONDITIONS: Premenstrual Syndrome; Uterus; Hemorrhage, Preclimacteric or Premenopausal
Keywords: Edema; Depression; Hot Flashes; Anxiety; Irritability; PMS
MeSH Terms: conditions — Premenstrual Syndrome; Hemorrhage; Edema; Depression; Hot Flashes; Anxiety Disorders | interventions — hypericin

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- GAMALINE® + HIPERICIN® 25-44 years old (Experimental): Fertile women 24-44 years old with PMS symptoms
  Interventions: Drug: GAMALINE® + HIPERICIN®
- GAMALINE® 25-44 years old (Active Comparator): Fertile women 24-44 years old with PMS symptoms
  Interventions: Drug: GAMALINE®
- GAMALINE® + HIPERICIN® 45-55 years old (Experimental): Climacteric women with PMS symptoms
  Interventions: Drug: GAMALINE® + HIPERICIN®
- GAMALINE® 45-55 years old (Active Comparator): Climacteric women with PMS symptoms
  Interventions: Drug: GAMALINE®

INTERVENTIONS:
Drug: GAMALINE® + HIPERICIN® — GAMALINE® 900mg + HIPERICIN 300mg T0 = 2 soft caps of each / day (1st month) T1-T6 = 1 soft caps of each / day (2nd - 6th month)
  Other Names: GAMALINE® BATCH 8663A0 MS 1.1860.0061.002-9; HIPERICIN® BATCH 867911 MS 1.1860.0003.003-0
  Arms: GAMALINE® + HIPERICIN® 25-44 years old; GAMALINE® + HIPERICIN® 45-55 years old
Drug: GAMALINE® — GAMALINE® 900mg T0= 2 soft caps / day (1st month) T1-T6 = 1 soft caps / day (2nd - 6th month)
  Other Names: GAMALINE® BATCH 8663A0 MS 1.1860.0061.002-9
  Arms: GAMALINE® 25-44 years old; GAMALINE® 45-55 years old

SUMMARY:
2 phytomedicines already in the market: GAMALINE® for premenstrual syndrome and HIPERICIN® as antidepressant will be prescribed together for treating women with Premenstrual Syndrome (PMS) symptoms and vasomotor problems for checking the advantage compared to the GAMALINE® prescription alone.

DETAILED DESCRIPTION:
Test with 2 female groups: 25-44 years old (reproductive age) and 45-55 years old (climacteric premenopausal age) complaining about all symptoms related with premenstrual syndrome.

ELIGIBILITY:
Inclusion Criteria:

* fertile women between 25-44 years old
* climacteric women between 45-55 years old

Exclusion Criteria:

* inferior age to 25 years old
* superior age to 55 years old
* post-menopausal
* under hormone therapy
* thyroid disease
* under psychiatric therapy or medication
* history for allergies and/or hypersensitivity to any component
* breast feeding or pregnancy
* no knowledge for writing and/or reading

Ages: 25 Years to 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 240 (Estimated)
Dates: Start 2012-03; Primary Completion 2012-10 (Estimated); Study Completion 2012-12 (Estimated)

PRIMARY OUTCOMES:
PMS calendar | 240 days
  Evaluation will run daily during the 240 days, comparing the results before treatment [60 days (T-2) and 30 days (T-1)]. Starting point (T0) treatment/under prescription, till 180 days treatment (T6).
LAB Tests | T0 T1 and T6
  Blood sample tests before T0 (all arms), after T1 (30 days only for experimental group) and end of T6 (after 180 days of prescription for all arms)

SECONDARY OUTCOMES:
WHOQOL | 06 months
  WHOQOL will be evaluated at T-2 and T6 where T-2 is at the first interview after inclusion and T6 is at the end point of treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Carla Vanin, MD MSc PhD, Principal Investigator — UFCSPA-Universidade Federal de Ciências da Saúde de Porto Alegre; Karla F Deud José, PharmD PhD, Study Chair — Phytopharm Consulting Brazil
Locations (1):
- Ambulatório de Ginecologia e Obstetrícia ISCMPA, Porto Alegre, Rio Grande do Sul, Brazil